CLINICAL TRIAL: NCT00060463
Title: Increased Access to Emergency Contraceptive Pills
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1R01HD039907 (NIH)
Record Dates: First submitted 2003-05-06; First posted 2003-05-07 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2004-10

CONDITIONS: Pregnancy; Sexually Transmitted Diseases
Keywords: Emergency contraceptive pills; Pregnancy; Sexually transmitted infection; Chlamydia; Gonorrhea; Trichomonas; Contraception
MeSH Terms: conditions — Sexually Transmitted Diseases; Chlamydia Infections; Gonorrhea; Trichomonas Infections

INTERVENTIONS:
Behavioral: Increased access to emergency contraceptive pills

SUMMARY:
This study will evaluate the effect of easy access to emergency contraceptive pills (ECPs) on the rates of pregnancy and sexually transmitted infections (STIs).

DETAILED DESCRIPTION:
ECPs are a back-up contraceptive method indicated for prevention of pregnancy after sexual intercourse if a primary contraceptive method fails or is not used. This trial will determine how increased access to ECPs affects the probability of pregnancy and three STIs. The STIs tested in the study are chlamydia, gonorrhea, and trichomonas. The trial will also evaluate how ready access to ECPs influences contraceptive or STI-prevention behaviors, particularly use of ECPs themselves, use of condoms, and use of other contraceptive methods.

The trial will be conducted among about 1,490 young women in the United States at high risk for pregnancy and STIs. Sexually active women aged 14 to 24 years who use barrier methods of contraception, oral contraceptive pills, or no contraception will be enrolled. Each woman will be randomly assigned to either an Advance Provision group or a Standard Care group. In the Advance Provision group, women will be given a supply of ECPs free of charge to keep at home in case of need. In the Standard Care group, women will be counseled about ECPs and invited to come to the clinic to obtain them at usual clinic charges when necessary.

Participants will be seen for follow-up at Months 6 and 12. At each visit, participants will be asked about pregnancies, STIs, sexual activity, self-assessed STI and pregnancy risk, and use of ECPs and other contraceptive methods. A specimen will be obtained for chlamydia, gonorrhea, and trichomonas testing.

ELIGIBILITY:
Inclusion Criteria

* Sexual intercourse with a male partner at least twice in the month prior to study entry
* Does not desire pregnancy within 1 year of study entry
* 6 weeks since the end of her last pregnancy and has had at least one menstrual period since resolution of her last pregnancy
* Literate in English or Spanish

Exclusion Criteria

* Surgically sterilized or intends to become sterilized within 1 year of study entry
* Intrauterine device or a hormonal implant in place or intends to have one inserted within 1 year of study entry
* Received an injection of a long-term contraceptive hormone (such as depot-medroxyprogesterone acetate) within 6 months of study entry or intends to receive one within 1 year of study entry
* Intends to use Lunelle, the vaginal contraceptive ring, or the contraceptive patch for contraception within 1 year of study entry
* Intends to use partners' vasectomy as her method of contraception within 1 year of study entry
* Pregnant or breastfeeding
* Known or suspected infertility
* Previously participated in this study
* Planning to move out of the study area within 1 year of study entry
* Currently participating in another research study that would interfere with the conduct of this study

Ages: 14 Years to 24 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 1490
Dates: Start 2002-10; Study Completion 2005-10

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Planned Parenthood Mar Monte / University of California at San Francisco, Reno, Nevada
  - Planned Parenthood of Central North Carolina, Durham, North Carolina

REFERENCES:
- [Derived] Weaver MA, Raymond EG, Baecher L. Attitude and behavior effects in a randomized trial of increased access to emergency contraception. Obstet Gynecol. 2009 Jan;113(1):107-116. doi: 10.1097/AOG.0b013e318190c0fe. PMID 19104366
- [Derived] Raymond EG, Stewart F, Weaver M, Monteith C, Van Der Pol B. Impact of increased access to emergency contraceptive pills: a randomized controlled trial. Obstet Gynecol. 2006 Nov;108(5):1098-106. doi: 10.1097/01.AOG.0000235708.91572.db. PMID 17077230